CLINICAL TRIAL: NCT06359366
Title: The Effect of Perineal Massage Combined With Hip Joint Training on Pelvic Floor Function
Brief Title: Perineal Massage Combined With Hip Joint Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Principal Investigator, Zonglian Guo, nurse, Shenzhen Hospital of Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ShenzhenH-guo
Record Dates: First submitted 2024-04-01; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: when the participants are enrolled in this study, they will be allocated to groups randomly by an independent researcher and sign the consent form. The care providers will not know the outcomes of this study, they just provide treatment for pregnant women; therefore, the care providers could be masked. an independent investigator will send a questionnaire to the participant, and the investigator does not know the intervention participants received; thus they could be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): perineal massage combined hip joint training
  Interventions: Procedure: perineal massage combined hip joint training
- comparison arm (No Intervention): Routine antenatal examination combined self-exercise

INTERVENTIONS:
Procedure: perineal massage combined hip joint training — pregnant women take the lithotomy position, disinfect the vulva, and wear sterile gloves. Then thumbs, forefingers, and middle fingers dip massage oil to do a 2 minutes pressurized dilatation massage from inside to outside gently to loosen the fascia. Then rest 30s. All steps need to be repeated 2 to 3 times. When the pregnant women feel a slight sense of acidity and tingling sensation disappears, researchers sterilize the perineal body again. left side pelvic floor receives the same intervention as right. The whole process takes 15-20min, 5 times a week until delivery. Additionally, while using the pelvic floor fascia manipulation, pregnant women are instructed to perform specific movements of internal and external hip rotation, adduction and abduction, upward and downward.
  Arms: intervention arm

SUMMARY:
The goal of this clinical trial is to learn if perineal massage combined with hip joint training works to improve pelvic function (urinary incontinence, constipation and hip motion) in pregnant women. The main questions it aims to answer are:

Does the perineal massage combined with hip joint training lower the prevalence of participants who have urinary incontinence and constipation? Does the perineal massage combined with hip joint training improve the flexibility of the hip joint? Researchers will compare an intervention (perineal massage combined with hip joint training) to a comparison(regular training and treatment) to see if the intervention (perineal massage combined with hip joint training) works to improve pelvic function.

Participants will:

receive the intervention (perineal massage combined with hip joint training ) or regular training and treatment fifth a week at 36 weeks gestation before participants receive first-time intervention, they complete Demographic sociological , ICI-Q-LF, Wexner constipation and hip motion questionnaires

DETAILED DESCRIPTION:
Women experience varying degrees of damage to the female reproductive and urinary muscle groups during pregnancy and delivery, which can lead to a series of pelvic floor disorders, for example, pelvic organ prolapse (POP), urinary incontinence(UI), chronic constipation (CC) and other syndrome, reducing the quality of life.

This study examined the effect of perineal massage combined with hip joint training on pelvic floor function, especially on UI, CC and hip motion. This is a parallel randomised control trial. The researchers will recruit participants from the obstetrics outpatient ward. Pregnant women attending the maternity clinic who met the inclusion and exclusion criteria will be randomly selected and sign informed consent, then the enrolled population was randomly assigned to each group using sealed envelopes.

The intervention group will receive perineal massage combined with hip joint training; the comparison group will receive regular training.

The primary outcome is the ICI-Q-LF score; Wexner constipation score; and the secondary outcome is hip motion.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnant women
* primipara;
* signed informed consent voluntarily
* 36 weeks gestation;
* no pregnancy complication

Exclusion Criteria:

* pluripara;
* multiple pregnancies;
* pregnant women with mental or cognitive disabilities;
* scarred uterus;
* pelvic surgery history;
* urinary incontinence before pregnancy history;
* obstipation before pregnancy history

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-04-10 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
pelvic floor function(constipation) | the outcomes will be assessed at 1.before the first time intervention at 36 gestational age. 2.receive intervention 10 times during two weeks(5 times/week). the results will reported through study completion, an average 3 months.
  using the Wexner Constipation Scoring System (lowest score, 0; Highest score, 30, contain 8 questions) to assess the outcomes of constipation. total score greater than 15 indicates constipation.the higher the score, the more difficult it is to defecate.
pelvic floor function (urinary incontinence score) | the outcomes will be assessed at 1.before the first time intervention at 36 gestational age. 2.receive intervention 10 times during two weeks(5 times/week). the results will reported through study completion, an average 3 months.
  using the ICI-Q-SF (containing 4 questions) to assess the degree of urinary incontinence. the higher the score, the worse the incontinence.

SECONDARY OUTCOMES:
hip motion | the outcomes will be assessed at 1.before the first time intervention at 36 gestational age. 2.receive intervention 10 times during two weeks(5 times/week). the results will reported through study completion, an average 3 months.
  The standard human range of motion scale(hip motion scale). Hip motion was measured under different exercise types.

CONTACTS AND LOCATIONS:
Overall Officials: wenjuan wang, master, Principal Investigator — matron

IPD SHARING:
Plan to Share IPD: Yes
study protocol could be share with others
Supporting Information: Study Protocol
Time Frame: after the paper has been published
Access Criteria: the detail in clinicaltrial.gov

REFERENCES:
- [Background] Jaekel AK, Kirschner-Hermanns R, Knupfer SC. [Diagnostic testing of female urinary incontinence: dos and dont's]. Aktuelle Urol. 2021 Jun;52(3):237-244. doi: 10.1055/a-1492-5287. Epub 2021 May 21. German. PMID 34020505
- [Background] Wang X,Li YJ,Deng ML.et al.Analysis of prevalence and risk factors of pelvic floor dysfunction in pregnant women[J].Nursing Research,2012,26(18):1636-1638
- [Background] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735
- [Background] Walker GJ, Gunasekera P. Pelvic organ prolapse and incontinence in developing countries: review of prevalence and risk factors. Int Urogynecol J. 2011 Feb;22(2):127-35. doi: 10.1007/s00192-010-1215-0. Epub 2010 Jul 9. PMID 20617303
- [Background] Cong X. Construction of evidence-based practice plan for postpartum pelvic floor rehabilitation management [D]. Beijing University of Chinese Medicine, 2024.
- [Background] Glazener C, Elders A, MacArthur C, Lancashire RJ, Herbison P, Hagen S, Dean N, Bain C, Toozs-Hobson P, Richardson K, McDonald A, McPherson G, Wilson D; ProLong Study Group. Childbirth and prolapse: long-term associations with the symptoms and objective measurement of pelvic organ prolapse. BJOG. 2013 Jan;120(2):161-168. doi: 10.1111/1471-0528.12075. Epub 2012 Nov 27. PMID 23190018